CLINICAL TRIAL: NCT04555057
Title: The Effects of Personalized Music Therapy to Reduce Patient Anxiety for Surgery on Patient-doctor Relationship and Patient Satisfaction
Brief Title: Music and Surgery Associated With Relationship and Satisfaction
Acronym: MARS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yohan Joo, Principal Investigator, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-1243
Record Dates: First submitted 2020-09-09; First posted 2020-09-18 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Music therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music therapy group (Experimental): One day before surgery, the participants of music therapy group choose the music they want to listen in the operating room. The total playing time of the selected music is recommended between 5 and 10 minutes.
  On the day of surgery, after entering the operating room, listen to personally selected music through the speaker. After the music is over, start anesthesia induction.
  Interventions: Procedure: Music therapy
- Control group (No Intervention): The participants of control group wear earmuff to block noise after entering the operating room until induction of anesthesia. All other treatments proceed as conventional treatments.

INTERVENTIONS:
Procedure: Music therapy — Music selected according to the patient's individual preferences.
  Arms: Music therapy group

SUMMARY:
In this study, the investigators want to check whether it has a direct effect on the participants first, and secondly, whether it affects the relationship between the patient and the doctor or treatment satisfaction, by reducing the anxiety of patients before surgery through music therapy.

DETAILED DESCRIPTION:
Patients often experience anxiety before surgery. They feel anxious for a number of reasons, such as worrying about the state of the disease they are diagnosed with, discomfort about the unfamiliar hospital environment, whether the operation is safe or it will be painful after surgery. In particular, anxiety related to surgery increases as the date and time of surgery approaches, and is most heightened just before surgery.

Persistent anxiety can lead to depression by triggering negative emotions, may also contribute to low compliance with overall treatment, and leading to low quality of life (QoL).

For this reason, various alternative treatments have been attempted to reduce the patient's stress, and music therapy is one of them. Music therapy can significantly reduce anxiety in patients before surgery. In addition, through many attempts so far, the possibility of affecting pain or quality of life after surgery has been confirmed. However, the results of studies are still inconsistent and evidence is not clear about the additional effects that can be obtained through patient anxiety reduction. Therefore, more earnest and practical research is required on additional effects and utilization through music therapy.

The investigators realized the possibility that listening to music to a patient before anesthesia in an operating room could not only reduce anxiety for the patient, but also provide an opportunity to improve the relationship with the doctor. Listening to music in the operating room is an impressive experience for the patient, and it can be an opportunity to make a positive impression on the medical staff who prepared it. This has the potential to improve the relationship between patients and doctors who need to continue to meet for additional treatment in the future.

According to a study by H. Beesley et al., in 40% of patients after breast reconstruction surgery, there was a difference between the satisfaction of the surgery and the cosmetic evaluation of the medical staff, and the relationship between the patient and the medical staff was evaluated to have an effect on this. A good relationship with a doctor or medical staff can lead to high satisfaction in patients with a low beauty score, and conversely, a poor relationship with a medical staff can lead to low satisfaction. This can be considered the possibility that if the patient-doctor relationship is improved through music therapy, the patient's satisfaction with surgery or treatment can also be increased.

The investigators will see how much anxiety can be reduced by listening to pre-operative music to patients. In addition, Researchers will evaluate the depth of the relationship between the patient and the doctor and find out whether there is a correlation with the patient's satisfaction with surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient with breast cancer
* Patients scheduled for surgery under general anesthesia

Exclusion Criteria:

* Patients with serious mental illness accompanied by cognitive impairment that makes voluntary independent judgment or social life impossible
* Patients with hearing impairment that makes it impossible to listen to music
* Patients with distant metastasis confirmed and performed as a palliative surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety scale | Change between anxiety scales on of about 15 minutes from immediately after entering the operating room to just before induction of anesthesia.
  An 11-point Numeric rating scale based on patient statements with 0 point for no anxiety and 10 for extreme anxiety.

SECONDARY OUTCOMES:
Changes in anxiety scale over time | Changes in the anxiety scale at 4 time points from the evening before surgery to immediately after entering the operating room on the day of surgery, immediately before induction of anesthesia, and 2 days after surgery.
  An 11-point Numeric rating scale based on patient statements with 0 point for no anxiety and 10 for extreme anxiety.
Changes in anxiety scale II | Changes in the anxiety scale from the evening before surgery to 2 days after surgery.
  Anxiety scale measured using Generalized Anxiety Disorder 7-item (GAD-7) scale. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
  The measurement of anxiety scale in the operating room has no choice but to be measured with the Numeric rating scale(NRS) stated by the patient due to time constraints. However, since the NRS score can be different for each individual, we intend to compensate for errors by measuring and comparing NRS and GAD-7 together on the day before and 2 days after surgery.
Patient-Doctor Depth-of-Relationship Scale(PDDR) | The PDDR score measured at 2 days after surgery.
  A single overall depth-of-relationship score can be calculated, which ranges from 0 (no relationship) to 32 (very strong relationship).
Satisfaction for surgery | The questionnaire about satisfaction is measured 2 days after surgery and 2 weeks after surgery.
  An 11-point scores measured through the questionnaire range from 0 (if not satisfied at all) to 10 (very satisfied).

OTHER OUTCOMES:
The participant's baseline depression score. | This score is measured at the evening before surgery.
  Measurement of patient baseline depression using Center for Epidemiologic Studies Depression Scale (CES-D). Possible range of scores is zero to 60, with the higher scores indicating the presence of more symptomatology.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palmer JB, Lane D, Mayo D, Schluchter M, Leeming R. Effects of Music Therapy on Anesthesia Requirements and Anxiety in Women Undergoing Ambulatory Breast Surgery for Cancer Diagnosis and Treatment: A Randomized Controlled Trial. J Clin Oncol. 2015 Oct 1;33(28):3162-8. doi: 10.1200/JCO.2014.59.6049. Epub 2015 Aug 17. PMID 26282640
- [Background] Bradt J, Dileo C, Magill L, Teague A. Music interventions for improving psychological and physical outcomes in cancer patients. Cochrane Database Syst Rev. 2016 Aug 15;(8):CD006911. doi: 10.1002/14651858.CD006911.pub3. PMID 27524661
- [Background] Beesley H, Ullmer H, Holcombe C, Salmon P. How patients evaluate breast reconstruction after mastectomy, and why their evaluation often differs from that of their clinicians. J Plast Reconstr Aesthet Surg. 2012 Aug;65(8):1064-71. doi: 10.1016/j.bjps.2012.03.005. Epub 2012 Apr 3. PMID 22475685
- [Background] Ridd MJ, Lewis G, Peters TJ, Salisbury C. Patient-doctor depth-of-relationship scale: development and validation. Ann Fam Med. 2011 Nov-Dec;9(6):538-45. doi: 10.1370/afm.1322. PMID 22084265
- [Background] Bayrak A, Sagiroglu G, Copuroglu E. Effects of Preoperative Anxiety on Intraoperative Hemodynamics and Postoperative Pain. J Coll Physicians Surg Pak. 2019 Sep;29(9):868-873. doi: 10.29271/jcpsp.2019.09.868. PMID 31455484